CLINICAL TRIAL: NCT01053624
Title: Concomitant Tracheostomy and Lung Resection in Patient With Low Postoperative Pulmonary Function
Brief Title: Concomitant Tracheostomy and Lung Resection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0064
Record Dates: First submitted 2010-01-05; First posted 2010-01-21 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Lung Cancer
Keywords: Tracheostomy and thoracic surgery; postoperative complications; pulmonary surgical procedures; respiratory failure
MeSH Terms: conditions — Lung Neoplasms; Postoperative Complications; Respiratory Insufficiency | interventions — Tracheostomy

INTERVENTIONS:
Procedure: Tracheostomy — This protocol has been design to determine if tracheostomy performed immediately after lung operation (i.e. concomitant tracheotomy) could improve the postoperative outcome of high risk patients. We hypothesized that concomitant tracheotomy could reduce the length of mechanical ventilation and the number of respiratory complications

SUMMARY:
This protocol has been designed to determine if tracheostomy performed immediately after lung operation (i.e. concomitant tracheotomy) could improve the postoperative outcome of high risk patients. We hypothesized that concomitant tracheotomy could reduce the length of mechanical ventilation and the number of respiratory complications.

DETAILED DESCRIPTION:
Background: Respiratory failure after lung resection is a major complication. Several studies suggest that low predictive postoperative pulmonary function is a predictive factor of mechanical ventilation (MV). In critically ill patients requiring MV, early tracheostomy may shorten the duration of MV and length of stay in intensive care.

Study objective: To determine whether concomitant tracheostomy (CT) would decrease the length of MV and improves outcome in patient with predictive postoperative forced expiratory volume in 1 second (FEV1ppo) < 50%. We call CT a tracheostomy performed immediately after the lung resection under the same general anesthesia.

Method: An open monocentric randomized controlled trial has been design. Inclusion and exclusion criteria are mentioned below. FEV1ppo will be calculated by the mean of the scintigraphic method for pneumonectomy and by the mean of the number of resected segments for lobectomy and segmentectomy. Randomization will be made the day before the operation. The procedure will be an open surgical tracheostomy. A daily data base will be completed from randomization until discharge. The primary and secondary criteria are mentioned below.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 79 years old
* preoperative diagnosis of suspected lung cancer
* patient considered operable according to the guidelines
* 30% < postoperative predicted FEV1 < 50%
* informed consent obtained by patient

Exclusion Criteria:

* - age less than 18 and more than 79
* pregnant woman
* preoperative tracheostomy
* postoperative vocal cord paralysis
* postoperative diaphragmatic paralysis (except for pneumonectomy)
* neuromuscular disorders
* previous pharyngeal or laryngeal surgery
* anatomical deformity of the neck making risky a tracheostomy
* consent refusal

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2001-10; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
number of mechanical ventilation days after operation until discharge | 2 months

SECONDARY OUTCOMES:
60 days mortality rate | 2 months
ICU length of stay | 2 months
hospital length of stay | 2 months
cumulative incidence of postoperative respiratory complications defined as pneumonia, re-ventilation, atelectasis needing fiberbronchoscopy, non cardiogenic pulmonary edema, air leakage >7 days, broncho-pleural fistula, pulmonary embolism, empyema | 2 months
cumulative incidence of postoperative cardiac complications defined as arrythmia needed treatment, cardiac failure needing inotrop drug, acute coronary stroke | 2 months
laryngeal and tracheal complications | 2 months
general complications | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Filaire, MD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Filaire M, Tardy MM, Richard R, Naamee A, Chadeyras JB, Da Costa V, Bailly P, Eisenmann N, Pereira B, Merle P, Galvaing G. Prophylactic tracheotomy and lung cancer resection in patient with low predictive pulmonary function: a randomized clinical trials. Chin Clin Oncol. 2015 Dec;4(4):40. doi: 10.3978/j.issn.2304-3865.2015.11.05. PMID 26730752